CLINICAL TRIAL: NCT04927728
Title: The Application of a Mental Practice Protocol to Increase the Functional Recovery of the Hemiparetic Upper Extremity in the Acute Inpatient Rehabilitation Setting
Brief Title: The Application of a Mental Practice Protocol in the Acute Inpatient Rehabilitation Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adventist HealthCare (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdventistHC
Record Dates: First submitted 2021-06-01; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: mental practice; stroke; upper extremity; hemiparesis; rehabilitation interventions
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Audio MP (Experimental): Participants of the audio mental practice (MP) group will complete MP via audio-guided multisensory cues of one of four tasks: (1) wiping a table (2) picking up a cup (3) brushing hair and/or (4) turning the page of a book. The assigned motor task is based upon the functional abilities of the patient. MP will be performed followed by physical practice of the same task with a research therapist 3x/week and independent MP 2 days/week. Each audio recording consists of 20 repetitions of the task.
  Interventions: Other: Mental Practice
- Video MP (Experimental): Participants of the video mental practice (MP) group will complete MP via video-guided multisensory cues of one of four tasks: (1) wiping a table (2) picking up a cup (3) brushing hair and/or (4) turning the page of a book. The assigned motor task is based upon the functional abilities of the patient. MP will be performed followed by physical practice of the same task with a research therapist 3x/week and independent MP 2 days/week. Each audio recording consists of 20 repetitions of the task.
  Interventions: Other: Mental Practice
- Repetitive-Task Practice (Experimental): Participants of the repetitive-task practice group will complete repetitive practice of one of four tasks: (1) wiping a table (2) picking up a cup (3) brushing hair and/or (4) turning the page of a book. The assigned motor task is based upon the functional abilities of the patient. MP will be performed followed by physical practice of the same task with a research therapist 3x/week and independent MP 2 days/week. Each participant completed at least 20 repetitions of the task.
  Interventions: Other: Repetitive-Task Practice
- Traditional Therapy (Active Comparator): The control group received traditional occupational therapy stroke rehabilitation.
  Interventions: Other: Traditional Therapy

INTERVENTIONS:
Other: Mental Practice — MP is the cognitive rehearsal of a motor task without physical movement, with the intent to improve motor performance. Mental practice can be completed via audio or video recording, visual prompts, written instructions, self-initiated or recorded pictures.
  Other Names: Mental Imagery; Motor Imagery
  Arms: Audio MP; Video MP
Other: Repetitive-Task Practice — Repetitive-Task Practice is the repetitive rehearsal of a motor task with the intent to improve motor performance.
  Other Names: Repetitive-Task Specific Practice
  Arms: Repetitive-Task Practice
Other: Traditional Therapy — Traditional therapy includes traditional interventions completed in occupational therapy for patients following a stroke. These interventions include but are not limited to, range of motion, weight-bearing, massage, modalities, self-care training, and transfer training.
  Arms: Traditional Therapy

SUMMARY:
The purpose of this randomized controlled trial is to compare the effect of audio-guided mental practice (MP) and video-guided MP on the impairment and functional abilities of upper extremity (UE) hemiparesis following a stroke. Participants are recruited from Adventist Healthcare Rehabilitation Hospital. All participants must be less than one-month post-stroke with moderate UE hemiparesis. Eligible participants are randomly assigned to an experimental group, (MP or repetitive-task practice (RTP)), or the control group.

The MP groups will perform either audio-guided MP or video-guided MP, five days a week, with 20 repetitions of the following tasks: wiping a table, picking up a cup, brushing hair, and turning the pages of a book. The RTP group physically performed the same tasks. The control group received traditional stroke rehabilitation.

The investigators hypothesize that video MP will have greater improvements in UE impairments and functional abilities than audio MP, RTP, and/or traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of stroke
* Less than one-month post-stroke
* Hemiparesis of one upper extremity
* Moderate upper extremity impairment

Exclusion Criteria:

* History of prior stroke
* Comorbidities (severe neurological, orthopedic, rheumatoid, or cardiac impairments)
* Severe spasticity
* Severe cognitive impairments
* Inability to perform mental imagery
* Severe aphasia based on speech therapist evaluation
* Low English proficiency
* Severe pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment-Upper Extremity Portion (FMA-UE) (Measuring pre/post intervention change) | Within 3 days of admission and within 3 days prior to discharge
  The Fugl Meyer Assessment-upper extremity(FMA-UE) portion will be administered to measure the impairment of the upper extremity. Upper extremity movements are rated on 3-point ordinal scale where 0= unable to perform, 1= performs partially, 2= performs fully. Cumulative scores range from 0-66 where a lower score indicates increased impairment.
Wolf Motor Function Test (WMFT) (Measuring pre/post intervention change) | Within 3 days of admission and within 3 days prior to discharge
  The Wolf Motor Function Test (WMFT) is used to measure the functional abilities of the UE. 15 tasks are performed including six timed joint-segment movements and eight timed integrative functional movements. Tasks are rated on a 6-point ordinal scale where 0= does not attempt to 5=movement appears to be normal. Timed and functional ability scores are calculated to indicate the functional abilities of the UE.

CONTACTS AND LOCATIONS:
Locations (1):
- Adventist Healthcare Rehabilitation, Rockville, Maryland, United States